CLINICAL TRIAL: NCT00723762
Title: Valproic Acid-associated Hypoalbuminemia in Medically Fragile Pediatric and Young Adult Patients in a Long Term Care Facility Part 1: Potential Mechanism for Decreased Albumin Synthesis
Brief Title: Valproic Acid-associated Hypoalbuminemia in Medically Fragile Patients
Status: Completed | Type: Observational
Sponsor: Akron Children's Hospital (Other)
Responsible Party: Michael Reed, Pharm.D., Akron Children's Hospital
Other Study IDs: Valproic Acid-Albumin
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Last update posted 2011-03-10 (Estimated); Status verified 2011-03

CONDITIONS: Hypoalbuminemia
Keywords: Valproic acid; Urea cycle; Ornithine; Valproate; Side effect
MeSH Terms: conditions — Hypoalbuminemia | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Control
Biospecimen Retention: Samples Without DNA — Serum and urine samples from patients receiving VPA.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Resident of Hattie Larlham long-term care facility receiving VPA
  Interventions: Procedure: Specimen collection
- 2: Control AED patients will be recruited based on similar AED regimens excluding VPA, length of time on AED (number of months to >1 year), age, and gender; one control patient per VPA patient.
- 3: Control non-AED patients will be recruited based on age and gender; one control patient per VPA patient.

INTERVENTIONS:
Procedure: Specimen collection — A blood sample and a spot urine sample will be obtained from all eligible patients receiving VPA at the start of the study.
  Groups: 1

SUMMARY:
The purpose of this study is to investigate potential mechanisms of valproic acid-associated low serum albumin in medically fragile pediatric and young adult epileptic patients of a long-term care facility.

DETAILED DESCRIPTION:
Valproic acid (VPA) is a long-chain fatty acid frequently used as an antiepileptic agent in pediatric and adult seizure patients. Other adverse effects that have been associated with VPA use include hepatic steatosis, altered mitochondrial function and decreased concentrations of serum proteins. The exact mechanism or mechanisms by which VPA induces these associated adverse drug effects are not fully understood though multiple theories have been postulated including impaired vesicle transport within the hepatocyte, inhibition of hepatic synthetic metabolic pathways and renal protein loss. Decreased serum albumin concentrations with concomitant VPA use have been identified in multiple studies. Albumin synthesis is sensitive to tryptophan concentrations (other amino acids are also able to stimulate albumin synthesis), oncotic pressure near the synthetic site, and energy supply while albumin release from the hepatocyte is sensitive to intrahepatocellular potassium concentrations. Based on available literature, VPA appears to inhibit an enzyme(s) either directly or indirectly involved with albumin synthesis or albumin gene expression. VPA is known to inhibit the urea cycle, including patients with ornithine-transcarbamylase (OTC) deficiency, possibly by inhibiting mitochondrial carbamoyl-phosphate synthase. Oratz et al discussed the potential correlation between the urea cycle and albumin synthesis identified after the administration of various amino acids increased both albumin and urea synthesis. Ornithine is an intermediate amino acid within the urea cycle and it is also a precursor to polyamines which have been shown to increase the degree of aggregation of polysomes, responsible for protein synthesis, bound to the endoplasmic reticulum. Thus, VPA may indirectly inhibit protein synthesis by interfering with the urea cycle leading to decreased ornithine concentrations and subsequently a decrease in polyamine concentrations and a decrease in the number of bound polysomes resulting in alterations in albumin synthesis and release. The purpose of this study is to investigate potential mechanisms of VPA-associated hypoalbuminemia in medically fragile pediatric and young adult epileptic patients of a long-term care facility.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Hattie Larlham long-term care facility receiving VPA for > 3 months at the start of the study
* Resident of Hattie Larlham long-term care facility matched to a resident receiving VPA for > 3 month based on concomitant AED, length of time on AED, age, and gender
* Resident of Hattie Larlham long-term care facility not receiving AED matched to a resident receiving VPA for > 3 month based on age and gender

Exclusion Criteria:

* Received albumin products within the past 1 month
* Receiving VPA for < 3 months or discontinuation of VPA therapy within the past four weeks
* Medical need for specific protein supplementation
* Diagnosed with protein-losing nephropathy or enteropathy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Medically fragile residents of the Hattie Larlham Long Term Care Facilit.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be serum albumin concentrations at baseline in the patients receiving VPA. | Baseline

SECONDARY OUTCOMES:
Secondary outcome variables will include serum amino acid concentrations, total protein, AST, ALT, alkaline phosphatase, ammonia, BUN, and sCr and urine albumin, protein, and urea. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Michael Reed, PharmD, Principal Investigator — Akron Children's Hospital Research Center; Martha Blackford, PharmD, Study Chair — Akron Children's Hospital; Richard Grossberg, MD, Study Chair — Hattie Larlham
Locations (1):
- Hattie Larlham Center for Children with Disabilities, Mantua, Ohio, United States

REFERENCES:
- [Background] Attilakos A, Voudris KA, Katsarou E, Prassouli A, Mastroyianni S, Garoufi A. Transient decrease in serum albumin concentrations in epileptic children treated with sodium valproate monotherapy. Clin Neuropharmacol. 2007 May-Jun;30(3):145-9. doi: 10.1097/wnf.0b013e3180318a99. PMID 17545749
- [Background] Hauser E, Seidl R, Freilinger M, Male C, Herkner K. Hematologic manifestations and impaired liver synthetic function during valproate monotherapy. Brain Dev. 1996 Mar-Apr;18(2):105-9. doi: 10.1016/0387-7604(95)00139-5. PMID 8733899
- [Background] Rugino TA, Janvier YM, Baunach JM, Bilat CA. Hypoalbuminemia with valproic acid administration. Pediatr Neurol. 2003 Nov;29(5):440-4. doi: 10.1016/s0887-8994(03)00310-2. PMID 14684241
- [Background] Oratz M, Rothschild MA, Schreiber SS, Burks A, Mongelli J, Matarese B. The role of the urea cycle and polyamines in albumin synthesis. Hepatology. 1983 Jul-Aug;3(4):567-71. doi: 10.1002/hep.1840030415. PMID 6407956
- [Background] Karikas GA, Schulpis KH, Bartzeliotou A, Karakonstantakis T, Georgala S, Kanavaki I, Demetriou E, Papassotiriou I. Lipids, lipoproteins, apolipoproteins, selected trace elements and minerals in the serum of children on valproic acid monotherapy. Basic Clin Pharmacol Toxicol. 2006 Jun;98(6):599-603. doi: 10.1111/j.1742-7843.2006.pto_402.x. PMID 16700824
- [Background] Castro-Gago M, Rodrigo-Saez E, Novo-Rodriguez I, Camina MF, Rodriguez-Segade S. Hyperaminoacidemia in epileptic children treated with valproic acid. Childs Nerv Syst. 1990 Dec;6(8):434-6. doi: 10.1007/BF00302087. PMID 2095300